CLINICAL TRIAL: NCT06002646
Title: Clinical and Radiographic Evaluation of Diode and Er:Cr;YSGG Lasers as an Alternative to Formocresol and Sodium Hypochlorite for Pulpotomy Technique in Primary Molars - Randomized Controlled Clinical Trial
Brief Title: Lasers as an Alternative to Formocresol and Sodium Hypochlorite Medicaments in Pulpotomy Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Wasan Adil, Principal investigator, University of Sulaimani
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: USaimani; Registration No.: 159/23 (Other: College of Dentistry/ University of Sulaimani)
Record Dates: First submitted 2023-08-01; First posted 2023-08-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pulp Disease, Dental; Pulp Mummification
MeSH Terms: conditions — Dental Pulp Diseases; Dental Pulp Necrosis | interventions — formocresol; Sodium Hypochlorite; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This randomized double blinded clinical trial in which both the participants(patients) and the investigator don't know about which type of treatment groups will be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- first group (Group A) (Active Comparator): using a 1:5 dilution of Buckley's FC (SSA, Produits Dentaires, Switzerland). A sterile cotton pellet will be moistened with a 1:5 concentration formocresol and it will be placed on the pulp stumps for 5 minutes for achieving hemostasis before being covered with MTA. If hemostasis will not be achieved after 5 minutes, it will presume that the pulp tissue in the canal was infected, and the tooth will be removed from the research
  Interventions: Drug: Formocresol
- second group (Group B) (Experimental): using 3% NaOCl(Tahno-dent, Greece) A sterile cotton pellet will be moistened with a 3% NaOCl and it will be placed on the pulp chamber for 5 minutes for achieving hemostasis before being covered with MTA
  Interventions: Drug: Sodium Hypochlorite Solution
- third group (Group C) (Experimental): In this group hemostasis will be achieved by exposure to diode laser (Biolase, epic X) of 940 nm. The laser energy will be introduced into the canal orifice through a 300 µm optical fiber at 2 W, in a contact mode with continuous mode CW(According to the user manual('EpicX_CAN_UM.pdf', no date) for 1 second at each orifice for three times to achieve complete hemostasis. During laser application patients, operator and assistant will use protective eye shields according to the safety measures of the device user manual.
  Interventions: Device: Diode laser
- fourth group (Group D) (Experimental): Irradiation of the floor of the pulp chamber with Er,Cr:YSGG laser 2790 nm (Waterlase MD, Biolase) at a Power of 1.5 w, Frequency of 50 Hz, mode S (soft tissue mode) , 20%air and no water with a gold handpiece and Tip type MZ6, for 10 sec.(According to the manufacturer manual iPlus™ software copyright ©2016 BIOLASE, Inc.)('WaterLase-iPlus-UM.pdf', no date). In which a fixed char layer should be formed over the pulpal tissue of the canals orifices. During laser application patients, operator and assistant will use protective eye shields according to the safety measures of the device user manual.
  Interventions: Device: Er,Cr:YSGG laser

INTERVENTIONS:
Drug: Formocresol — Hemostasis of pulpal tissue in primary teeth pulpotomy techniques with Formocresol solution
  Other Names: Buckley's solution
  Arms: first group (Group A)
Drug: Sodium Hypochlorite Solution — Hemostasis of pulpal tissue in primary teeth pulpotomy techniques with 3% Sodium Hypochlorite Solution.
  Other Names: NaOCl
  Arms: second group (Group B)
Device: Diode laser — Hemostasis of pulpal tissue in primary teeth pulpotomy techniques with 940 nm diode laser.
  Arms: third group (Group C)
Device: Er,Cr:YSGG laser — Hemostasis of pulpal tissue in primary teeth pulpotomy techniques with 2790nm Er,Cr:YSGG laser.
  Other Names: Erbium, Chromium: Yttrium-Scandium-Gallium-Garnet laser
  Arms: fourth group (Group D)

SUMMARY:
The goal of this clinical trial is to evaluate the dental lasers as an alternative of chemical medicaments used in the pulpotomy procedures. The main question it aims to answer is:

• Lasers pulpotomies are a viable alternative to the standard Formocresol and Sodium Hypochlorite medicaments.

All participants groups (Formocresol, Sodium Hypochlorite, Diode and Er:Cr;YSGG lasers) for pulpotomy procedure will follow the same clinical protocol, except for the techniques that will be used for hemostasis of the pulpotomies which either will be achieved by Formocresol or Sodium Hypochlorite solutions or by Diode or Erbium lasers.

DETAILED DESCRIPTION:
All the selected treatment groups (Formocresol, Sodium Hypochlorite, Diode and Er:Cr;YSGG lasers) will follow the same clinical protocol, except for the techniques that will be used for hemostasis of the pulpotomies:

1. Using 2 percent lidocaine with 1: 100,000 epinephrine as a local anesthetic.
2. Isolation of the teeth with a rubber dam.
3. Using a diamond round #440 bur in a high-speed hand piece with water cooling to eliminate caries and expose pulp chambers.
4. Using a spoon excavator to remove the coronal pulp.
5. Achieving the hemostasis by:

I. In first group (Group A): using a 1:5 dilution of Buckley's FC solution. A sterile cotton pellet will be moistened with a 1:5 concentration formocresol and it will be placed on the pulp stumps for 5 minutes for achieving hemostasis before being covered with MTA. If hemostasis will not be achieved after 5 minutes, it will presume that the pulp tissue in the canal was infected, and the tooth will be removed from the research.

II. In the second group (Group B): using 3% NaOCl. A sterile cotton pellet will be moistened with a 3% NaOCl and it will be placed on the pulp chamber for 5 minutes for achieving hemostasis before being covered with MTA.

III. In the third group (Group C): In this group hemostasis will be achieved by exposure to diode laser of 940 nm. The laser energy will be introduced into the canal orifice through a 300 µm optical fiber at 2 W, in a contact mode with continuous mode CW (According to the user manual) for 1 second at each orifice for three times to achieve complete hemostasis. During laser application patients, operator and assistant will use protective eye shields according to the safety measures of the device user manual.

IV. In the fourth group (Group D): Irradiation of the floor of the pulp chamber with Er,Cr:YSGG laser 2790 nm ) at a Power of 1.5 w, Frequency of 50 Hz, mode S (soft tissue mode) , 20%air and no water with a gold handpiece and Tip type MZ6, for 10 sec.(According to the manufacturer manual iPlus™ software copyright ©2016 BIOLASE, Inc.). In which a fixed char layer should be formed over the pulpal tissue of the canals orifices. During laser application patients, operator and assistant will use protective eye shields according to the safety measures of the device user manual.

1. Then covering the surface with a 2 mm layer of MTA
2. The final restoration will be completed in all the four groups, stainless steel crown will be placed as the final restorative material with a well-fitting marginal adaption and glass ionomer cement(GC company).

ELIGIBILITY:
Inclusion Criteria:

* Deep carious lesions present in primary molars.
* No history of spontaneous or persistent pain.
* Lack of clinical evidence of pulpal degeneration, such as pain on percussion, history of swelling or sinus tracts.
* Restorable teeth following completion of the procedure.
* Absence of radiographic signs and symptoms of pulpal degeneration.
* Following pulpal amputation, hemostasis could be easily achievable.

Exclusion Criteria:

* Uncooperative children.
* Children with medically compromised disease.
* Presence of radiographical signs and symptoms of pulpal degeneration.
* Physiologic root resorption is more than one-third.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical and radiographical success rate of pulpotomy procedure of FC, and NaOCl techniques and two different types of lasers Diode and Erbium Cr,YSGG lasers | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Wasan Adil Fadhil, Sulaymaniyah, Iraq

REFERENCES:
- [Derived] Fadhil WA, Noori AJ. Clinical and Radiographic Evaluation of Diode and Er,Cr:YSGG Lasers as an Alternative to Formocresol and Sodium Hypochlorite for Pulpotomy Techniques in Primary Molars: A Randomized Controlled Clinical Trial. Cureus. 2024 Jul 31;16(7):e65902. doi: 10.7759/cureus.65902. eCollection 2024 Jul. PMID 39219956